CLINICAL TRIAL: NCT01904162
Title: Determination of the Effect of Age and Gender on the Pharmacokinetics and Tolerability of a Single Dose of Finafloxacin-HCL in Healthy Volunteers
Brief Title: Effect of Age and Gender on the PK and Tolerability of Finafloxacin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MerLion Pharmaceuticals GmbH (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FINA-005; AA83723 (Other: CRO, MDS Pharma Services Protocol ID)
Record Dates: First submitted 2013-07-17; First posted 2013-07-22 (Estimated); Last update posted 2024-03-13 (Actual); Status verified 2013-07

CONDITIONS: Pharmacokinetic and Tolerability of Finafloxacin
MeSH Terms: interventions — finafloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- healthy young adult males (Experimental): healthy young adult males receiving 400 mg finafloxacin single dose
  Interventions: Drug: 400 mg finafloxacin (2 x 200 mg tablets)
- healthy young adult females (Experimental): healthy young adult females receiving 400 mg finafloxacin single dose
  Interventions: Drug: 400 mg finafloxacin (2 x 200 mg tablets)
- healthy elderly adult males (Experimental): healthy elderly adult males receiving 400 mg finafloxacin single dose
  Interventions: Drug: 400 mg finafloxacin (2 x 200 mg tablets)
- healthy elderly adult females (Experimental): healthy elderly adult females receiving 400 mg finafloxacin single dose
  Interventions: Drug: 400 mg finafloxacin (2 x 200 mg tablets)

INTERVENTIONS:
Drug: 400 mg finafloxacin (2 x 200 mg tablets)

SUMMARY:
Previous clinical studies have indicated that finafloxacin is well-tolerated with few treatment-related adverse events. As a part of the clinical development of finafloxacin, other PK studies are required to determine the effect of other variables on the PK profile of finafloxacin. This study aims to determine the effect of age and gender on the pharmacokinetic profile of finafloxacin.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male and/or female, 18 to 35 years of age (inclusive), or 65 years or over(≥ 65 years).
* Body mass index (BMI) ≥ 18 and ≤ 30 kg/m2.
* No clinically significant abnormal findings, as judged by the Principal Investigator (PI), on the physical examination, ECG, medical history, or clinical laboratory results during screening.
* Negative screen for human immunodeficiency virus (HIV), hepatitis B, C and/or positive hepatitis B surface antigen (HBsAg), and anti-Hepatitis C virus (HCV) antibodies.
* Females of childbearing potential were either sexually inactive (abstinent) for 14 days prior to the first dose and throughout the study or were using one of the following acceptable birth control methods:

  1. Surgically sterile (bilateral tubal ligation, hysterectomy, bilateral oophorectomy) for a minimum of 6 months.
  2. Intrauterine device (IUD) in place for at least 3 months.
  3. Barrier methods (condom and diaphragm) plus spermicide for at least 14 days prior to the first dose and throughout the study.
  4. Surgical sterilization of the partner (vasectomy for 6 months minimum).
  5. Hormonal contraceptives for at least 3 months prior to the first dose of the study and throughout the study.
* Females of non-childbearing potential were either postmenopausal for at least 2 consecutive years prior to Day 1, with a follicle-stimulating hormone (FSH) level > 40 IU/mL or had undergone one of the following sterilization procedures at least 6 months prior to Day 1:

  1. Bilateral tubal ligation.
  2. Hysterectomy.
  3. Hysterectomy with unilateral or bilateral oophorectomy.
  4. Bilateral oophorectomy.
* Male subjects were either sexually inactive (abstinent) or using a barrier method for 14 days prior to the first dose and throughout the study.
* In addition, male subjects and female subjects of childbearing potential were advised to remain sexually inactive or to keep the same birth control method for at least 30 days in the case of females and 90 days in the case of males, following the last dose. Male subjects were additionally advised not to donate sperm for 90 days following the last dose.
* Was able to understand and willing to sign an ICF.

Exclusion Criteria:

* Subject with psychiatric, neurological, or behavioral disorders that may have interfered with the conduct or interpretation of the study.
* Subject with a history or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, or hematological disorders that were capable of significantly altering the absorption, metabolism, or elimination of drugs, or were considered a risk with the study medication or could have interfered with the interpretation of data.
* Subject who had an abnormality in the 12-lead ECG that, in the opinion of the PI, increased the risks associated with participating in the study.
* Subject with clinically relevant abnormal laboratory data or vital signs at screening, or any abnormal laboratory value which, in the opinion of the PI, could have interfered with the assessment of safety.
* Subject with exposure to any investigational drug within 30 days prior to screening.
* Subject with a known hypersensitivity or other contraindication to the use of fluoroquinolones.
* Subject with a history of tendon rupture or tendonitis.
* Subject who received corticosteroid therapy in the 4 weeks prior to study drug administration.
* Subject with prior participation in a finafloxacin investigational study.
* Subject who had current diagnosis or known history of drug and/or alcohol abuse.
* Subject who smoked > 10 cigarettes per day and was unable or unwilling to refrain from nicotine during study confinement.
* Subject who received any drugs known to strongly inhibit or induce any of the enzymes within the cytochrome P-450 (CYP) system within 30 days prior to the first dose.
* Subject who had exposure to any medication (with the exception of hormone replacement therapy [HRT] for the elderly subjects), including over-the-counter (OTC) medications, 7 days prior to dosing.
* Subject who had exposure to antacid medication 24 hours prior to study drug administration until collection of the last PK sample.
* Subject who had consumed grapefruit 10 days prior to study drug administration until collection of the last PK sample.
* Subject with any clinically significant illness 3 months before the study.
* Subject who had donated blood or plasma during the previous 56 days prior to dosing.
* Subject who was unlikely to comply with the clinical study protocol.
* Subject who was a member of the clinical site or Sponsor personnel or their immediate family, defined as spouse, parent, sibling, child, grandparent, or grandchild.
* Any other condition that, in the opinion of the PI, precluded participation in the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-02; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic | Day 1
  The primary PK endpoints of the study were the 90% confidence interval (CI) for the ratio of the population geometric means of the PK parameters AUC0-t, AUC0-24, AUC0-inf, and Cmax in plasma and the 90% CI for the ratio of the population geometric means of the PK parameters CumAe0-24 and Rmax in urine.

SECONDARY OUTCOMES:
Safety and tolerability | Day 1
  1. The number and severity of treatment-emergent adverse events (TEAEs) following single doses of finafloxacin for each population in the study
  2. Changes from baseline for each population for safety clinical laboratory parameters, electrocardiographs, vital signs, and physical examinations

CONTACTS AND LOCATIONS:
Locations (1):
- Celerion (formerly MDS Pharmaservices), Tempe, Arizona, United States